CLINICAL TRIAL: NCT00101790
Title: A Pilot Trial of IV Pamidronate for Low Back Pain
Brief Title: A Pilot Trial of Intravenous (IV) Pamidronate for Low Back Pain
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Marco Pappagallo, MD;, The Mount Sinai Medical Center, New York, New York, United States, 10029
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: R01NS044845 (NIH)
Record Dates: First submitted 2005-01-13; First posted 2005-01-14 (Estimated); Last update posted 2010-01-07 (Estimated); Status verified 2010-01

CONDITIONS: Low Back Pain
Keywords: low back pain; pamidronate
MeSH Terms: conditions — Low Back Pain | interventions — Pamidronate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator)
  Interventions: Drug: pamidronate

INTERVENTIONS:
Drug: pamidronate — There will be four study groups, each with 7 subjects randomly assigned to pamidronate and 4 to placebo. The groups will occur in succession, not parallel. The dosage for group 1 will be 30 mg , 60 mg for group 2, and 90 mg for group 3. Group 4 will receive 2 treatments of 90mg IV pamidronate or placebo.

SUMMARY:
The purpose of this study is to determine the test dose of pamidronate for treatment of low back pain in terms of safety, tolerability, and pain relief.

DETAILED DESCRIPTION:
Chronic low back pain-an enormous clinical problem which affects large segments of populations throughout the world-causes disability and loss of productivity, and leads to enormous costs in healthcare resources. Efforts to find relatively non-invasive therapies for individuals suffering from this problem are important.

The main objective of this single-center, double-blind study is to determine the optimal dosing regimen-based on safety, tolerability, and pain relief- which should be used in planning a future, large-scale, clinical study to clarify conclusively whether chronic low back pain, unrelated to cancer, can be treated with pamidronate.

Forty-four persons will be recruited for participation. There will be four study groups, each with 7 subjects randomly assigned to pamidronate and 4 to placebo. The dosage for the pamidronate participants will be 30 mg of pamidronate for the first group, 60 mg for the second group, and 90 mg for the third group. Members of the fourth group will receive 2 treatments of 90mg IV pamidronate or placebo.

In this study, scientists also hope to find out if the effectiveness of pamidronate can be predicted with bone scans (a procedure used to see bone inflammation or injuries to the bone), and if improvement in performance of daily tasks is related to the amount of pamidronate a participant receives and to improvement in pain intensity, and to evaluate patient satisfaction with the pamidronate treatments.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, 21 years of age or older
* Having mechanical low back pain (LBP) that is predominantly axial, i.e., subjects with low back pain with proximal radiation (above the knee), or subjects with low back pain with distal radiation of pain (below the knee), only if their low back pain component is 50% or more than their leg pain component. This pain will have been present for at least 3 months, with a minimum, average pain score of 4 on a 0-10 numeric rating scale [NRS; a score of 4 is associated with pain of "moderate" intensity, and its use as a cutoff value is supported by the clinical relevance of similar scores found by others.
* MRI evidence of multiple level disc degeneration and vertebral changes consistent with the diagnosis of degenerative disc disease or spondylotic disease of the spine.
* Being capable of reading at a sixth-grade level.

Exclusion Criteria:

* Prior back surgery
* Compression fracture(s)
* Cancer that can be a possible cause of the back pain
* MRI evidence of frank disk herniation or any other abnormality or pathology (other than disc degeneration and vertebral changes consistent with the diagnosis of degenerative disc disease or spondylotic disease of the spine) regarding the probable cause of the patient's spinal pain; for example, arachnoiditis, moderate to severe spinal canal stenosis, lateral recess stenosis, congenital malformation of the spine, spinal nerve tumor, etc.
* Clinical diagnosis of relevant radiculopathic / neuropathic pain with leg pain, i.e., subjects with low back pain with distal radiation of pain (below the knee) if their leg pain component is more than 50% than their back pain component, or subjects with back pain with neurological deficits consistent with lumbosacral radiculopathy (upon examination)
* Presumptive compression of a spinal nerve root or fracture of a pars interarticularis (3) Spondylolisthesis (greater than grade one or more than 4 mm)
* A history of hypocalcemia
* Abnormal lab values:

  * A baseline value for liver function that is 5% or more above the upper normal limit
  * Upon the first laboratory screen, we will exclude anyone whose creatinine level is more than 5% outside the normal range. Then, of those who have acceptable creatinine levels, we will exclude anyone with a glomerular filtration rate (GFR) that is less than 60. The GFR will be calculated according to Levey et al.
  * The principal investigator will use his judgment regarding excluding any individual with other abnormal lab values.
* A history of significant cardiac, hematological, renal, hepatic, metabolic, endocrinological, or neurological disease
* An allergy to bisphosphonates
* Leukopenia or thrombocytopenia
* Being pregnant or nursing
* Diagnosis of painful polyneuropathy, e.g., painful diabetic neuropathy
* Psychotic symptoms. Dr. Barry Snow, the study consulting psychologist, will train study staff to recognize these symptoms.
* Alcohol abuse or illicit drug use
* Receiving Worker's Compensation, or having a pending Worker's Compensation claim
* Being blind, deaf, or mute, or having a physical or mental handicap that impedes administration of instruments that will provide outcome data
* Weighing less than 45 kg (this is rare for an adult)
* Subjects who are suicidal according to the Beck Depression Inventory, or score 26 and above on the Beck Depression Inventory will be excluded from the study.
* Prior pamidronate treatment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2003-09; Primary Completion 2010-06 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Best dose of pamidronate to be tested in a future large-scale study for treatment of low back pain. Criteria for best dose relate to safety/efficacy of the tested doses in this pilot trial | Length of study

CONTACTS AND LOCATIONS:
Overall Officials: Marco Pappagallo, MD, Principal Investigator — The Mount Sinai Medical Center
Locations (1):
- The Mount Sinai Medical Center, New York, New York, United States